CLINICAL TRIAL: NCT05075486
Title: Collaborative Quality Improvement to Reduce Mortality or Severe Intracranial Hemorrhage in Neonatal Extracorporeal Life Support in China
Brief Title: Quality Improvement to Reduce Mortality or Severe Intracranial Hemorrhage in Neonatal Extracorporeal Life Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Chinese Neonatal Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQI-RMSIH
Record Dates: First submitted 2021-09-06; First posted 2021-10-12 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Extracorporeal Life Support; Extracorporeal Membrane Oxygenation; Quality Improvement; Intracranial Hemorrhage; Mortality; Neonate
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Intervention Model Description: This is a pre- and post- interventional study in one group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Group who recieve collaborative quality improvement during study period.
  Interventions: Behavioral: Collaborative quality improvement

INTERVENTIONS:
Behavioral: Collaborative quality improvement — Hospitals will receive standardized center-specific ECLS data report with benchmarking to feedback on their performance. Evidence-based potential better practice list will be established as a reference for all hospitals. During the intervention period, the hospitals will receive training in collaborative quality improvement method and then develop, implement, and document evidence-based practice changes to reduce adverse outcomes of neonatal ECLS treatment. Compliance with practice changes and neonatal outcomes will be monitored. All hospitals will have access to implementation support and collaborative activities.

SUMMARY:
This is a three-year pre- and post- interventional study to assess the effectiveness of collaborative quality improvement interventions on reducing mortality and severe intracranial hemorrhage (ICH) for neonates receiving extracorporeal life support (ECLS) in China.

DETAILED DESCRIPTION:
This is a three-year pre- and post- interventional study from 2022 to 2024. The population of this study will be all neonates who receive ECLS support within 28 days of life in the participating hospitals of Chinese Neonatal Extracorporeal Life Support Registry (Chi-NELS). The intervention will be collaborative quality improvement interventions for each of the participating hospital. Detailed interventions include standardized ECLS data feedback and benchmark, establishment of potential better practice list, training on quality improvement, implementation of practice change using plan-do-study-action cycles, report and monitor of practice change and collaborative learning. The first year will be pre-intervention baseline period and serves as the control period. Collaborative quality improvement interventions will be introduced from the start of the second year and the second and third years will be the intervention period. The primary outcome, which is the incidence of mortality or severe ICH of the third year, will be compared to that of the baseline year.

ELIGIBILITY:
Inclusion Criteria:

* ≤28 days of life
* receive ECLS support

Exclusion Criteria:

* Infants with severe congenital anomalies
* Infants with pre-ECLS ICH

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality or severe intracranial hemorrhage (ICH) before discharge | From admission to discharge or death, an average of 3 months
  It is a binary variable (1/0). The variable would be set into "1", if death or severe ICH occurred

SECONDARY OUTCOMES:
Mortality | From admission to discharge or death, an average of 3 months
  Incidence of infants who died during hospitalization
Incidence of severe ICH | From admission to discharge or death, an average of 3 months
  Proportion of infants who have severe ICH during hospitalization
Incidence of successful decannulation of extracorporeal life support | From admission to discharge or death, an average of 3 months
  Proportion of infants who removed from extracorporeal life support successfully
Incidences of ECLS related complications | From admission to discharge or death, an average of 3 months
  Complications include mechanical complications, hemorrhage (GI, cannulation site, surgical site), brain death, seizures, CNS diffuse ischemia, CNS infarction, renal failure, CPR required, cardiac arrhythmia, pneumothorax, pulmonary hemorrhage, hemolysis, limb ischemia, and infection. It is a binary variable (1/0). The variable would be set into "1", if any complication occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Cao, Principal Investigator — Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No